CLINICAL TRIAL: NCT04560153
Title: Interest of Karate Kata Practice on the Self-esteem of Patients Living With HIV
Acronym: KATACHRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier le Mans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CHM-2019/S10/05
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2020-09-24 (Actual); Status verified 2020-09

CONDITIONS: Patients Living With HIV
Keywords: HIV; KARATE KATA; SELF ESTEEM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patient living with HIV (Experimental)
  Interventions: Other: karate kata

INTERVENTIONS:
Other: karate kata — sessions of karate kata every week during 4 months

SUMMARY:
Since ancient times, physical and sports activity has been recognized as bringing many health benefits. Descriptive and interventional studies on physical activity are developing, demonstrating physical and psychological benefits for patients with various diseases.

Physical activity is effective in improving self-esteem in the general population. Good self-esteem allows for better autonomy to manage a chronic illness.

The benefit of physical activity in patients living with HIV has been the subject of several studies, notably outside France, and seems to improve the quality of life.

We hypothesize that sport, especially karate kata, could improve self-esteem in patients living with HIV, and represent another non-drug aid, in patients living with HIV.

ELIGIBILITY:
Inclusion Criteria:

* patient living with HIV
* Patient seen in the infectious diseases department of Le Mans hospital, during a consultation or day hospitalization for HIV follow-up
* Aged 18 years and older
* Patients able to understand and to give informed consent to participate in the study
* valid social security coverage
* written and signed informed consent by the patient and investigator

Exclusion Criteria:

* refusal to participate to the study
* pregnant or brest-feeding women
* person subject to a legal protection measure
* patient with psychiatric disease
* patient under legal protection
* medical contraindication to play karate kata

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Effect of karate kata training on self-esteem among patients living with HIV followed at the Le Mans hospital center | 4 months
  Change from Baseline at 4 months as assessed by Rosenberg's questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Du Mans, Le Mans, France

REFERENCES:
- [Derived] Grandiere Perez L, Duveau T, Lelong C, Dangeul F, Hitoto H, Blanchi S. Favorable effect of Karate Kata on self-esteem, anxiety and fatigue in people living with HIV. Psychol Health Med. 2025 Feb 28:1-12. doi: 10.1080/13548506.2025.2472050. Online ahead of print. PMID 40019027